CLINICAL TRIAL: NCT00085878
Title: A Phase I, Dose Escalation Study to Assess the Safety and Pharmacokinetics of SB- 485232 Administered as Daily Subcutaneous Injections in Adult Patients With Solid Tumors
Brief Title: Dose-Escalation Study Of SB-485232 Administered As Daily Subcutaneous Injections In Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 485232/002; 002
Record Dates: First submitted 2004-06-16; First posted 2004-06-18 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Solid Tumor Cancer
Keywords: IL-18; subcutaneous; pharmacokinetics; Phase 1
MeSH Terms: interventions — Interleukin-18

INTERVENTIONS:
Drug: SB-485232

SUMMARY:
This is a phase I, open-label, dose-escalation study of SB-485232. Subjects will receive SB-485232 administered as subcutaneous injections daily for 14 days. Dose escalation (enrollment into the next cohort) cannot occur until all three subjects have completed the previous cohort; 5 doses will be tested. An additional dosing regimen has been added to evaluate higher doses given twice weekly for 7 weeks. Therefore, the full evaluation period for each patient will extend out to approximately eleven weeks after the first day of SB-485232 dosing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of malignancy.
* Subjects with solid tumors must have locally advanced or metastatic disease at the time of enrollment.
* Measurable or evaluable disease that is refractory or resistant to standard therapy or for which there is no effective standard therapy.
* Predicted life expectancy of at least 12 weeks.
* Kinesin spindle protein (KPS) of greater than 70%.
* No chemotherapy, immunotherapy, hormonal therapy, or biological therapy for cancer, radiotherapy, or surgical procedures (except for minor surgical procedures) within 4 weeks before beginning treatment with SB-485232 (6 weeks for nitrosoureas and mitomycin C).
* Subjects must have recovered from toxicities (incurred as a result of previous therapy) sufficiently to be entered into a Phase I study.
* Provide written informed consent.
* Absence of anti-SB-485232 antibodies.
* Hemoglobin greater than or equal to 9 g/dL.
* Absolute neutrophil count greater than or equal to 1.5 X 109 /L.
* Platelet count greater than or equal to 100 X 109 /L.
* Partial thromboplastin time (PTT) and prothrombin time/international normalized ratio (PT/INR) within normal limits.
* Serum creatinine less than or equal to 1.5 mg/dL (135 µmol/L) or estimated creatinine clearance greater than 50 mL/min (calculated by the Cockcroft-Gault Formula).
* Total serum bilirubin less than or equal to 1.5 mg/dL.
* Aspartate transaminase (AST) and alanine transaminase (ALT) less than or equal to 3 X ULN.
* Sexually active males or females of reproductive capacity must use adequate contraception.
* For subjects with a history of coronary artery disease, stress test must be within normal limits.
* Subjects with a history of congestive heart failure, myocardial infarction or prior anthracycline chemotherapy must have a Multiple Gated Acquisition (MUGA) scan with a left ventricular ejection fraction of greater than 40%.

Exclusion Criteria:

* Women who are pregnant or are breast-feeding.
* Severe or uncontrolled infections requiring systemic antibiotic therapy.
* Any serious medical or psychiatric disorder that would interfere with subject safety or informed consent.
* Known leptomeningeal disease or evidence of prior or current metastatic brain disease.
* Receiving concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy.
* Receiving concurrent systemic steroids.
* History of ventricular arrhythmias requiring drug or device therapy.
* Any severe concurrent disease or condition, including significant autoimmune diseases, which in the judgment of the principal investigator, would make the subject inappropriate for study participation.
* Any unresolved or unstable serious toxicity from prior administration of another investigational drug.
* Any investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of SB-485232.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the study.
* Received prior treatment with SB-485232.
* Poor venous access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-01

PRIMARY OUTCOMES:
- Safety and tolerability endpoints will include evaluation of adverse events and changes in laboratory values and clinical variables from pre-dose values. | 11 Weeks

SECONDARY OUTCOMES:
- Biologically effective dose based. - Pharmacokinetic endpoints: AUC, Adverse Events, cmax, tmax, and t1/2. - Presence or absence of anti-SB-485232 antibodies. - Pharmacodynamic endpoints. - Radiographic tumor assessments. | 11 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania